CLINICAL TRIAL: NCT01894386
Title: An Open Label, Randomised, Four-Period Crossover, Single Dose Study in Healthy Volunteers to Evaluate the Pharmacokinetics of FF/UMEC/VI Combination Administered at Dose Levels 100/62.5/25 mcg and 100/125/25 mcg and in Comparison With FF/VI (100/25 mcg) and UMEC/VI (62.5/25 mcg).
Brief Title: Pharmacokinetic Study in Healthy Volunteers to Characterise the Exposure of Fluticasone Furoate (FF), Vilanterol (VI) and Umeclidinium (UMEC) at Two Different Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200587
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GW642444 (Vilanterol); GSK573719 (Umeclidinium); GW685698 (Fluticasone Furoate); pharmacokinetics; Healthy subjects
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental): Subjects will receive treatment A, B, C, D in each dosing periods 1, 2, 3, and 4 respectively (one per period). A - FF/UMEC/VI 400/500/100; B - FF/UMEC/VI 400/250/100; C - FF/VI 400/100; D - UMEC/VI 250/100
  Interventions: Drug: FF 400 mcg; Drug: UMEC 500 mcg; Drug: UMEC 250 mcg; Drug: VI 100 mcg
- Sequence 2 (Experimental): Subjects will receive treatment B, D, A, C in each dosing periods 1, 2, 3, and 4 respectively (one per period). A - FF/UMEC/VI 400/500/100; B - FF/UMEC/VI 400/250/100; C - FF/VI 400/100; D - UMEC/VI 250/100
  Interventions: Drug: FF 400 mcg; Drug: UMEC 500 mcg; Drug: UMEC 250 mcg; Drug: VI 100 mcg
- Sequence 3 (Experimental): Subjects will receive treatment C, A, D, B in each dosing periods 1, 2, 3, and 4 respectively (one per period). Subjects will receive treatment B, D, A, C in each dosing periods 1, 2, 3, and 4 respectively (one per period). A - FF/UMEC/VI 400/500/100; B - FF/UMEC/VI 400/250/100; C - FF/VI 400/100; D - UMEC/VI 250/100
  Interventions: Drug: FF 400 mcg; Drug: UMEC 500 mcg; Drug: UMEC 250 mcg; Drug: VI 100 mcg
- Sequence 4 (Experimental): Subjects will receive treatment D, C, B, A in each dosing periods 1, 2, 3, and 4 respectively (one per period). Subjects will receive treatment C, A, D, B in each dosing periods 1, 2, 3, and 4 respectively (one per period). Subjects will receive treatment B, D, A, C in each dosing periods 1, 2, 3, and 4 respectively (one per period). A - FF/UMEC/VI 400/500/100; B - FF/UMEC/VI 400/250/100; C - FF/VI 400/100; D - UMEC/VI 250/100
  Interventions: Drug: FF 400 mcg; Drug: UMEC 500 mcg; Drug: UMEC 250 mcg; Drug: VI 100 mcg

INTERVENTIONS:
Drug: FF 400 mcg — 100 mcg powder for inhalation delivered by Dry Powder Inhaler (DPI)
Drug: UMEC 500 mcg — 125 mcg powder for inhalation delivered by DPI
Drug: UMEC 250 mcg — 62.5 mcg powder for inhalation delivered by DPI
Drug: VI 100 mcg — 25 mcg powder for inhalation delivered by DPI

SUMMARY:
This study will evaluate the pharmacokinetics of FF, UMEC and VI administered from one inhaler (at two different strengths of UMEC (125 and 62.5microgram [mcg]) and FF/VI (ICS/LABA) and UMEC/VI (LAMA/LABA).

Subjects will receive each of the four treatments once, separated by a wash-out period of 7-21 days between doses in a four way crossover design. There will be 4 treatment periods in total. During each treatment period, subjects will attend the clinical unit on Day -1 for standard safety assessments in addition to familiarization with the inhaler. Each subject will remain resident in the unit until at least 24 hours after the dose given on Day 1. Following completion of all four treatment periods, a follow up visit will take place 7 to 21 days following the final dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

Safety

* Average Corrected QT Interval using Fridericia's formula (QTcF) <450 msec at screening.
* Forced Expiratory Volume in 1 second (FEV1) >=80% predicted and a FEV1/Forced Vital Capacity (FVC) ratio >=0.7 at screening.
* Alanine transaminase (ALT), alkaline phosphatase and bilirubin <=1.5x Upper Limit Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Population

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and lung function testing. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and GSK medical monitor consider the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures and outcome.
* Subjects who are current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of <=10 pack years. [number of pack years = (number of cigarettes per day /20) x number of years smoked]
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* A female subject is eligible to participate as follows: Non-childbearing potential, females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods and women of childbearing potential should have used one of the contraception methods.
* Body Mass Index (BMI) within the range 18.0-33.0 kg/m2 (inclusive).

Exclusion Criteria:

Safety

* Lactating or pregnant females as determined by positive serum or urine hCG test at screening or Day -1.
* A supine mean heart rate outside the range 40-90 beats per minute (bpm) at screening.

Hepatic Disease

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or a history of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.

Concurrent Disease

* History of respiratory disease (i.e. history of asthmatic symptoms) in the last 10 years.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening or a positive test for HIV.

Concurrent Medication

* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

Population

* A positive pre-study drug/alcohol screen at screening and Day -1.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer), or has had exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* The subject is unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and pummelos, exotic citrus fruits, grapefruit hybrids or any fruit juices containing these fruits from 7 days prior to the first dose of study medication and for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-07-15 (Actual); Primary Completion 2013-09-26 (Actual); Study Completion 2013-09-26 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetic (PK) Parameters as a measure of systemic exposure. | PK Blood samples will be collected at Predose, 3, 5, 7, 10, 15, 12, 15, 30, 45 minutes, 1hour, 1.5, 2, 4, 6, 8, 12, 24 hours post dose on Day 1 of each treatment period
  Area under the concentration time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)) (or Area under the concentration time curve from time zero (pre-dose) to last common time of quantifiable concentration within a subject across all treatments [AUC(0-t')] if AUC(0-infinity) cannot be determined) and maximum observed concentration (Cmax) for each individual component (UMEC will be dose-normalised) across treatment groups will be estimated using the following treatment ratios: FF/UMEC/VI 100mcg/125mcg /25mcg Versus, FF/UMEC/VI 100mcg /62.5mcg /25mcg
Systemic exposure of FF and UMEC and VI following single inhaled doses (four inhalations) of FF/UMEC/VI 100mcg /62.5mcg /25mcg compared with FF/VI 100mcg /25mcg and UMEC/VI 62.5mcg /25mcg | PK Blood samples will be collected at Day 1 Predose, 3, 5, 7, 10, 15, 12, 15, 30, 45 minutes, 1hour, 1.5, 2, 4, 6, 8, 12, 24 hours post dose.
  FF: FF/UMEC/VI versus FF/VI; UMEC: FF/UMEC/VI versus UMEC/VI; VI: FF/UMEC/VI versus FF/VI; VI: FF/UMEC/VI versus UMEC/VI

SECONDARY OUTCOMES:
Composite of PK Parameters. | PK Blood samples will be collected at Day 1 Predose, 3, 5, 7, 10, 15, 12, 15, 30, 45 minutes, 1hour, 1.5, 2, 4, 6, 8, 12, 24 hours post dose.
  Elimination half-life of a compound (t½) and Time after administration of a compound when the maximum plasma concentration is reached (tmax)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 200587 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200587?search=study&search_terms=200587#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 200587 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200587 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200587 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200587 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200587 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200587 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200587 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register